CLINICAL TRIAL: NCT03747094
Title: Fentanyl Versus Ketamine Supplementation for Prpofol Anesthesia During Balloon Insertion in Morbidly Obese Patients
Brief Title: Sedation of Morbidly Obese for Balloon Insertion
Acronym: SedBaloon
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, lecturer of anesthesia, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sedation for balloon insertion
Record Dates: First submitted 2018-11-13; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Fentanyl; Ketamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fentanyl group (Active Comparator)
  Interventions: Drug: Fentanyl
- Ketamine group (Experimental)
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Fentanyl — 0.5 mic/kg fentanyl will be given immediately before the procedure
  Arms: Fentanyl group
Drug: Ketamine — 0.25 mg ketamine will be administered immediately before the procedure
  Arms: Ketamine group

SUMMARY:
This prospective study will assess the value of different supplements to orpofol bases anesthesia in morbidly obes e patients scheduled for balloon insertion. Two common drugs will be added to propofol bases anesthesia;Ketamine or fentanyl. Effect on prpofol consumption, post-procedure recovery profile, and patient satisfaction will be the study objectives.

ELIGIBILITY:
Inclusion Criteria:

* morbid obese indicated for gastric balloon insertion

Exclusion Criteria:

- Refusal Hypersensitivity to any of the study drugs

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-03-20 (Estimated); Study Completion 2019-04-15 (Estimated)

PRIMARY OUTCOMES:
Propofol consumption (milligrams) | 24 hours after the endoscopy
  Dose of prpofol (mg/kg) required for sedation during gastric balloon insertion

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Manşūrah, Dkahleya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided